CLINICAL TRIAL: NCT03481595
Title: Improvement of Patient Satisfaction and Overall Outcomes Using HealthLoop to Manage the Episode of Care for THA and TKA Bundles
Brief Title: Improvement of Patient Satisfaction and Overall Outcomes Using HealthLoop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Accelero Health Partners, LLC (Other); Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Carlos Higuera-Rueda, Vice Chair for Quality and Patient Safety, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-1496
Record Dates: First submitted 2018-03-02; First posted 2018-03-29 (Actual); Results first posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Arthroplasty, Replacement, Knee; Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group A (No Intervention): Group A will receive standard, routine medical care. If you are randomized to standard, routine medical care you will need to communicate with your Doctor and clinical care team through conventional methods such as over the phone or through MyChart.
- Group B (Experimental): Group B will be asked to use the HealthLoop mobile application on their mobile device during the post-operative period in addition to standard, routine medical care. Patients randomized to use the Health Loop app will be able to communicate with their Doctor and clinical care team directly through the app. Patients will also participate in mobile and web-based surveys, receive reminders related to their healthcare, and receive information personalized to their treatment plan.
  Interventions: Device: HealthLoop mobile application

INTERVENTIONS:
Device: HealthLoop mobile application — Patients will utilize the HealthLoop mobile application on their mobile device during the post-operative period in addition to standard, routine medical care.
  Arms: Group B

SUMMARY:
The purpose of this study is to assess the usefulness and results of orthopedic patients having access to a cell phone App called HealthLoop to utilize during the postoperative time period, compared to patients who have the usual postoperative management. The researchers want to investigate whether there any differences in outcomes and satisfaction in patients and providers.

DETAILED DESCRIPTION:
The purpose of this study is to assess the usefulness and results of orthopedic patients having access to a cell phone App called HealthLoop to utilize during the postoperative time period, compared to patients who have the usual postoperative management. The researchers want to investigate whether there any differences in outcomes and satisfaction in patients and providers.

HealthLoop is a mobile-device application (cell phone App) that allows physicians to monitor for signs and symptoms of potential adverse events, and communicate with patients during the postoperative recovery process. The platform enables doctors to identify patients at risk of decline in the follow up period. Patients are engaged through mobile and web-based surveys, reminders, and information personalized to the patient's specific condition or treatment plan. Alerts are sent to physicians about patients who are at risk of treatment failures, complications, or hospital readmissions. Physicians are informed if patients are trending toward an adverse outcome based on the patient's responses.

Patients who choose to participate in this Research Study will be randomly assigned (like a flip of a coin) to one of two groups. Group A will receive standard, routine medical care. Group B will be asked to use the HealthLoop application on their mobile device during the post-operative period in addition to standard, routine medical care. Patients will not be able to choose which group they will be in.

ELIGIBILITY:
Inclusion Criteria:

* Primary total hip arthroplasty or total knee arthroplasty patient
* Personal or surrogate consent to participate
* Patient has internet access or mobile access with a valid email address at the time of enrollment

Exclusion Criteria:

* Staged arthroplasty procedure within 6 months of the index procedure
* Abandoned email address of record
* Less than 14 days until date of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Higuera, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B
Started | 146 | 148
Completed | 143 | 127
Not Completed | 3 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 143 | 127 | 270
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (9) | 65 (8) | 66 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 67 | 148
  Male | 62 | 60 | 122
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting a Problem Across al PPE-15 Domains
Description: 15-item patient experience questionnaire. Each response will be categorized as a problem or non-problem and reported as the percent of respondents reporting a problem, averaged across all PPE-15 domains.
Time Frame: 90 days after index surgery
Measure: Mean (Standard Deviation); unit: percent of participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 143 | 127
percent of participants | 12.6 (15.3) | 9.5 (13.2)

2. Secondary Outcome: Visual Analog Scale (VAS) for Patient Satisfaction
Description: Satisfaction measurement tool measured on a scale from 0-100 mm. Where 0 = not satisfied and 100 = entirely satisfied.
Time Frame: 90 days after index surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 143 | 127
units on a scale | 91.0 (17.3) | 91.0 (13.9)

3. Secondary Outcome: Length of Hospital Stay
Description: A count of the number of days the patient was admitted to the hospital after the index procedure prior to being discharged. Measured in days.
Time Frame: 90 days after index surgery
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group A | Group B
Number analyzed (Participants) | 143 | 127
days | 1.4 (0.9) | 1.2 (0.7)

4. Secondary Outcome: Number of Participants Discharged to Home
Description: Was the patient routinely discharged to home? Reported as yes or no.
Time Frame: 90 days after index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 143 | 127
Participants | 130 | 118

5. Secondary Outcome: Number Participants Who Were Readmitted to the Hospital
Description: A count of the number of hospital readmissions related to the index procedure within 90 days after the index procedure.
Time Frame: 90 days after index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 143 | 127
Participants | 9 | 9

6. Secondary Outcome: Number Participants Who Visited the Emergency Department
Description: A count of the number of emergency department visits related to the index procedure within 90 days after the index procedure.
Time Frame: 90 days after index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 143 | 127
Participants | 24 | 19

7. Secondary Outcome: Number Participants With 0, 1, 2, or 3+ Outpatient Visits
Description: A count of the number of outpatient follow-up visits with the surgical team related to the index procedure within 90 days after the index procedure.
Time Frame: 90 days after index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 143 | 127
Participants
  0 follow up visits | 0 | 2
  1 follow up visit | 21 | 17
  2 follow up visits | 76 | 61
  3 or more follow up visits | 46 | 47

8. Secondary Outcome: Number of Participants Who Made 0, 1, 2, or 3+ Telephone Calls to the Surgical Team
Description: A count of the number of telephone calls with the surgical team related to the index procedure within 90 days after the index procedure.
Time Frame: 90 days after index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 143 | 127
Participants
  0 phone encounters | 15 | 12
  1 phone encounter | 37 | 40
  2 phone encounters | 39 | 32
  3 or more phone encounters | 52 | 43

9. Secondary Outcome: Number of Participants Who Had a Reoperation
Description: A count of the number of reoperations related to the index procedure within 90 days after the index procedure.
Time Frame: 90 days after index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 143 | 127
Participants | 1 | 4

ADVERSE EVENTS:
Time Frame: 90 days following total knee or total hip arthroplasty
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/143 | 1/127
Serious Adverse Events (participants affected / at risk) | 11/143 | 14/127
Other Adverse Events (participants affected / at risk) | 12/143 | 10/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=143) | Group B (N=127)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Manipulation under anesthesia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Hyperkalemia (Endocrine disorders) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Effusions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Gastrointestinal bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Allergy (Immune system disorders) | 0 (0) | 1 (1)
Transverse myelitis (Nervous system disorders) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
GI distress (Gastrointestinal disorders) | 1 (1) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Suture abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Hiccups (hospitalized) (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=143) | Group B (N=127)
swelling (General disorders) | 2 (2) | 3 (3)
hypotension (General disorders) | 4 (4) | 4 (4)
UTI (Renal and urinary disorders) | 3 (3) | 3 (3)
nausea (General disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/95/NCT03481595/Prot_SAP_001.pdf